CLINICAL TRIAL: NCT02878382
Title: Efficacy of Calcipotriol Assisted MAL-PDT Versus Conventional MAL-PDT for Actinic Keratosis: a Randomized and Controlled Study
Brief Title: Potential Impact of Patient Vitamin D Status in AK Response to MAL-PDT
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luis Antonio Torezan, Assistant Professor of Dermatology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08/2016
Record Dates: First submitted 2016-08-10; First posted 2016-08-25 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Actinic Keratosis
Keywords: PDT; skin cancer; calcipotriol
MeSH Terms: conditions — Keratosis, Actinic; Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional MAL-PDT (Other): Conventional topical PDT with Methylaminolevulinate 16% in one half of the scalp with multiple AKs.
  Interventions: Other: Conventional MAL-PDT
- Calcipotriol assisted MAL-PDT (Other): Calcipotriol ointment 50 mcg/g applied once a day for 15 consecutive days in one half of the scalp, before Conventional topical PDT
  Interventions: Other: Calcipotriol assisted MAL-PDT

INTERVENTIONS:
Other: Conventional MAL-PDT — Curettage of lesions and application of MAl cream 16% for 90 minutes under occlusion followed by LED 635 nm illumination at 37 J/cm2 total dose
  Arms: Conventional MAL-PDT
Other: Calcipotriol assisted MAL-PDT — Calcipotriol 50 mcg/g for 15 days prior to PDT. Curettage of lesions and application of MAl cream 16% for 90 minutes under occlusion followed by LED 635 nm illumination at 37 J/cm2 total dose
  Arms: Calcipotriol assisted MAL-PDT

SUMMARY:
In topical photodynamic therapy (PDT) for non-melanoma skin cancers, a photosensitizing prodrug, 5-aminolaevulinic acid (ALA) or its methylated ester, methyl aminolevulinate (MAL), is converted to the endogenous photosensitizer protoporphyrinIX (PpIX).

Reduced response rates are observed in thicker skin lesions, which may be due to insufficient PpIX accumulation within the target tissue.

To enhance PpIX production,several physical and chemical pretreatments have been suggested. One of the chemical substances proposed to stimulate PpIX production is vitamin D because of its ability of being a keratinocyte pro-differentiating hormone.

Based on in vitro and in animal model studies, we propose to study the potential impact of patient vitamin D pre-treatment in AK response to MAL-PDT.

DETAILED DESCRIPTION:
A randomized, controlled Split -scalp study with Calcipotriol Assisted MAL-PDT versus conventional MAL-PDT for actinic keratosis (AK) is proposed.

Twenty patients ( male gender only) with symmetrically distributed multiple AK lesions on the scalp will be included. Patients must have at least five AKs per field to be eligible.

After simple randomization, one half of the scalp will be treated with Calcipotriol ointment 50 mcg/g (Daivonex, Leo Pharma, Denmark) for 15 consecutive days.

After this period, the entire scalp will be submitted to topical PDT with Methylaminolevulinate 16% (Metvix, Galderma France) under occlusion for 90 minutes and then, illuminated with a light source consisting of a Light Emitting Diode device (LED) at 635 nm ( Aktilite - Photocure, Norway). The total light dose will be 37J/cm2.

Immediately before and after illumination with LED, measurements of the fluorescence intensity will be taken in 3 isolated spots in both sides of the scalp with a spectroscopy deviceUSB 2000+ ( Ocean Optics ® - Dunedin, Fl, USA).

AK lesions will be counted and mapped by a dermatologist not involved in the study before and after 3 months.

All patients will be advised to apply sunscreens 50 + 3x/day for the following 7 days after the procedure.

A 0-10 Visual Analogue Scale (VAS) will be used to measure the pain intensity during the illumination.

Records will be taken after 90 days and compared between sides: side effects, AK lesion response and pain level intensity. Also, a long term follow up will be provided at 6 and 12 months after.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* at least six AKs per field

Exclusion Criteria:

* history of photosensitivity related disorders
* active infectious disease,
* immunosuppression
* laser or any cosmetic treatment in the previous 6 months
* other topical agents in the treatment area such as retinoids, 5-fluorouracil,imiquimod or diclofenac sodium in the previous 3 months
* allergy to MAL or excipients of the cream
* poor patient compliance.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Torezan, MD, Principal Investigator — Hospital das Clinicas FMUSP Sao Paulo
Locations (2):
- Brazil (2):
  - Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital Das Clinicas Universidade Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All twenty patients completed the 12 -month study. Patients were male, Fitzpatrick skin types I-III and mean age 73.8 years (range 54-89).
Units Other Than Participants: half scalp
Groups:
- Calcipotriol Assisted MAL-PDT: Calcipotriol + MAL-PDT half scalp
- Conventional MAL-PDT: MAL-PDT alone half scalp
Period: Overall Study
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Started | 20; 20 half scalp (total 20 patients.split-scalp: 20 split -scalp received CAL-PDT and the other 20 received C-PDT) | 20; 20 half scalp (otal 20 patients.split-scalp: 20 split -scalp received CAL-PDT and the other 20 received C-PDT)
Completed | 20; 20 half scalp | 20; 20 half scalp
Not Completed | 0; 0 half scalp | 0; 0 half scalp

BASELINE CHARACTERISTICS:
Population: 20 male patients were selected and enrolled in the study. The eligibility criteria were: male sex, minimum age of 50 years old, at least 6 AKs symmetrically distributed on the scalp, only AKs grades I and II and immunocompetent patients. To receive either Conventional PDT or CAL-PDT on the allocated side of the scalp (right or left)
Groups:
- All Participants: Conventional topical PDT with Methylaminolevulinate 16% in one half of the scalp with multiple AKs.
  Conventional MAL-PDT: Curettage of lesions and application of MAl cream 16% for 90 minutes under occlusion followed by LED 635 nm illumination at 37 J/cm2 total dose
  Calcipotriol ointment 50 mcg/g applied once a day for 15 consecutive days in one half of the scalp, before Conventional topical PDT Calcipotriol assisted MAL-PDT: Calcipotriol 50 mcg/g for 15 days prior to PDT. Curettage of lesions and application of MAl cream 16% for 90 minutes under occlusion followed by LED 635 nm illumination at 37 J/cm2 total dose
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20
number of AKs at baseline [Number; unit: number of lesions] — AKs were clinically divided in 2 categories: grade I and grade II, based on Olsen et al classification. Grade I is a thinner lesion. Grade II is a thicker lesion. Both types co-exist on the same patient and reflects the skin photodamage.
  number of lesions
    CAL-PDT side | 290
    Conventional PDT | 284
    CAL-PDT side grade I | 223
    CAL-PDT side grade II | 67
    Conventional PDT grade I | 222
    Conventional PDT grade II | 62

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Actinic Keratosis - Lesion Base Count.
Description: To compare the efficacy of topical PDT alone versus Calcipotriol assisted PDT for AKs on the scalp.
  The values in the data table represent the mean (+sd) number of lesions on each side at 3, 6 and 12 months post intervention.
  Lesion counts include lesions that have not been cleared and also newly emerged lesions ( if new lesions emerge on the treated field) At baseline: number of AKs was 290 on the CAL-PDT side and 284 on the conventional side.
Time Frame: Change from baseline, 90 days, 180 days and 12 months after the PDT
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Calcipotriol Assisted MAL-PDT: Calcipotriol 15 days before - once a day intervention: MAL-PDT plus curettage Illumination LED 635 nm 37J/cm2
- Conventional MAL-PDT: intervention: MAL-PDT plus curettage Illumination LED 635 nm 37J/cm2
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Number analyzed (Participants) | 20 | 20
lesions
  3 months outcome | 1.15 (0.99) | 2.65 (1.35)
  6 months outcome | 1.15 (0.93) | 2.60 (1.14)
  12 months outcome | 1.35 (1.04) | 3.20 (1.44)
Statistical Analysis 1: Comparison: Calcipotriol Assisted MAL-PDT vs Conventional MAL-PDT; Test type: Superiority; p < 0.001, Chi-squared — significance level of 5%; also, Fisher's exact test and Mann-Whtiney were used for comparing the other variables in the study

2. Primary Outcome: Percentage of Actinic Keratosis (AK) Lesions Cleared
Description: AK clearance after PDT and comparison between the sides The values in the data table represent the percentage of AK clearance on each side at 3, 6 and 12 months post intervention.
  At baseline: 290 on the CAL-PDT side and 284 on the conventional side.
Time Frame: Change from baseline, 90 days, 6 months and 12 months after PDT
Measure: Number; unit: percentage of lesions cleared
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Number analyzed (Participants) | 20 | 20
percentage of lesions cleared
  3 months outcome | 92.1 | 82
  6 months outcome | 92.1 | 81.7
  12 months outcome | 90.7 | 77.5

3. Secondary Outcome: Pain Scores Immediately Post Illumination
Description: Measurement of pain during LED illumination and comparison between the sides with a visual analogue scale (VAS), considering 0 as absence of pain and 10 as the most severe pain.
  At baseline, before the illumination, there is an absence of pain, which means Score 0 (zero) for all participants before the procedure.
  Pain is reffered during and after the illumination and measured with the VAS scale, reported by each patient.
Time Frame: immediately after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Number analyzed (Participants) | 20 | 20
units on a scale | 5.4 (1.4) | 4.0 (0.69)
Statistical Analysis 1: Comparison: Calcipotriol Assisted MAL-PDT vs Conventional MAL-PDT; Test type: Superiority; p = 0.001, Fisher Exact — significance level of 5%

4. Secondary Outcome: Change From Baseline in Fluorescence Intensity of PPIX
Description: Measurement of PPIX fluorescence on both sides of the scalp before and immediately after LED illumination PpIX fluorescence was measured in three different spot areas on the scalp before and immediately after PDT on each side.
  The measurements were taken noninvasively in the areas where PpIX fluorescence was more intense, with a handheld fluorescence photometer (USB 2000+ spectroscopy device; Ocean Optics, Dunedin, FL, U.S.A.). The photometer illuminates a circular skin area with a diameter of 1 cm with blue light (400-420 nm), matching the Soret band of PpIX at 405-420 nm. By measuring excitation wavelengths at 600- 700 nm, the corresponding red PpIX fluorescence intensity at 633 nm is detected. Measurements were taken in arbitrary units. The mean PpIX fluorescence value for each side was calculated before and after the treatment.
Time Frame: Baseline and 10 minutes after illumination
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Number analyzed (Participants) | 20 | 20
arbitrary units | 3422.85 (1775.19) | 2688.35 (1746.12)
Statistical Analysis 1: Comparison: Calcipotriol Assisted MAL-PDT vs Conventional MAL-PDT; Student's t-test or the Mann-Whitney test was used according to the assumption of normality of data for PpIX fluorescence intensity; Test type: Superiority; p = 0.048, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: side effects collected over 10 days
Description: During light exposure patients were asked to evaluate the intensity of pain using a visual analogue scale (VAS), considering 0 as absence of pain and 10 as the most severe pain. Local skin reactions (erythema, edema, pustules, crusts, erosions and ulcerations) were recorded as well as any systemic adverse events during treatment and after follow-up visits. Clinical assessments of the local skin reactions were performed on a pre-defined scale as: 0 = no reaction, + mild, ++ moderate, +++ severe
Arm/Group | Calcipotriol Assisted MAL-PDT | Conventional MAL-PDT
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 15/20 | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcipotriol Assisted MAL-PDT (N=20) | Conventional MAL-PDT (N=20)
local skin reactions (Skin and subcutaneous tissue disorders) | 15 (22) | 12 (20) — erythema, edema, crusts and pustules.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No